CLINICAL TRIAL: NCT04543734
Title: A Feasibility and Usability Study of HemoScreen Hematology Analyzer for Cancer Patients Receiving Chemo and Its Potential for Home Monitoring of Blood Values Before Chemotherapy
Brief Title: The Potential of HemoScreen for Monitoring Blood Values in Cancer Patients at Home
Status: Completed | Type: Observational
Sponsor: Niels Henrik Holländer (Other)
Responsible Party: Sponsor-Investigator, Niels Henrik Holländer, Chief physician, MD, Naestved Hospital
Organization: Naestved Hospital (Other)
Other Study IDs: Hem2020
Record Dates: First submitted 2020-08-24; First posted 2020-09-10 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: Cancer; Complete blood count; Point-of-care; HemoScreen
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HemoScreen hematology analyzer — The use of HemoScreen for self-testing of blood values

SUMMARY:
To keep cancer patients safe, whilst in chemo therapy, patients come into the hospital for multiple blood tests, in order to provide safe antineoplastic treatment and supportive care. Monitoring of relevant blood values (WBC white blood cell count, total and differentiated, ANC absolute neutrophil count, RBC red blood cell count, HGB hemoglobin and PLT platelets) is usually obtained by venipuncture by a health-care professional at the hospital.

HemoScreen is a POCT (point-of-care-technology) automated hematology analyzer that performs complete blood count (CBC) analysis from capillary or venous whole-blood samples. HemoScreen solution has not yet been used by patients to self-test blood cell count, but the investigators hypothesize that cancer patients on systemic anticancer therapy can perform a self-test at home using HemoScreen, and transfer the results to the hospital clinical team, to prevent wasted hospital journeys. This study aims to investigate the feasibility and usability of HemoScreen hematology analyzer for capillary self-testing of blood values in home for cancer patients receiving chemo.

The study consists of a quantitative and a qualitative part. The quantitative part is to compare blood values obtained by capillary self-testing using HemoScreen and venous blood values obtained on standard hospital equipment (Sysmex) in patients. The qualitative part will be observational studies and semi-structured interviews with patients as well as health professionals from the department of Clinical Oncology, as they perform a capillary blood test with HemoScreen themselves. Recruitment of participants will take place at the department of Clinical Oncology in Naestved.

This present study has two phases. The first phase (1) will investigate feasibility, usability and measurement properties of the HemoScreen CBC analyzer, when patients perform a capillary self-test in the outpatient clinic at Oncology supervised by trained personal. Furthermore, Healthcare professionals will test the capillary blood count method. Phase 1 will be conducted to insure that HemoScreen is safely used for capillary self-testing by patient before initiating phase 2, where the HemoScreen is being sent home with the patients for self-measure at home. In Phase 1, 10 cancer patients as well as 4-10 health professionals will be recruited. In phase 2, 33 cancer patients initiating a chemotherapy treatment will be recruited for testing in their home.

DETAILED DESCRIPTION:
Background In Denmark the specialty of clinical oncology, provides complex and high-risk medical treatment to patients diagnosed with solid malignancies. To keep patients safe, whilst in therapy (with a curative or palliative intend), patients come into the hospital for multiple blood tests, physical evaluation, registration and treatment of possibly life-threatening adverse effects, all in order to provide safe antineoplastic treatment and supportive care. A low neutrophil blood cell count (neutropenia) can be a dose-limiting toxicity of systemic anti-cancer therapy and can be life-threatening when complicated by sepsis. Neutrophil count is usually obtained by venipuncture by a health-care professional. Correspondingly this applies for the loss of blood production (anemia) and loss of production of blood platelets (thrombocytopenia).

Exploring new ways to closely monitor and treat future cancer patients aiming at increasing quality of life, as well as reducing the cost in hospital tests and admissions, must be given high priority.

HemoScreen is a POCT automated hematology analyzer that performs complete blood count (CBC) analysis from capillary or venous whole-blood samples, using a single use self-contained cartridge. The cartridge is preloaded with all required reagents. After analysis, the results are displayed and can be saved, printed, or exported to another digital system. The HemoScreen Analyzer provides 20 standard CBC parameters in approximately 6 minutes RBC, absolute WBC count, WBC 5-part differential and PLT.

The HemoScreen CBC was developed to be used by professionals and therefore, the HemoScreen solution has not yet been used by patients to self-test complete blood cell count.

The investigators hypothesize that cancer patients on systemic anticancer therapy can measure a home blood count using HemoScreen, record quantitative data and transfer the results to the hospital clinical team. Future intentions are to trial the use of the HemoScreen CBC analyzer to reduce frequency and severity of neutropenia, anemia and thrombocytopenia complications, prevent wasted hospital journeys and hospital resources, reduce non-elective hospital admissions and personalize delivery of anticancer treatment.

The HemoScreen CBC analyzer has shown rapid and accurate test results for both venous and capillary blood samples, when compared to standard measurement (Sysmex). Also in the lower range, relevant for monitoring and post chemotherapy treatment in cancer patients.

This present study has two phases. The first phase of this study (1) will investigate feasibility, usability and capillary measurement properties of the HemoScreen CBC analyzer, when patients self-test their blood cell count when in the outpatient clinic at Oncology and supervised by trained personal. Furthermore, Healthcare professionals will test the capillary blood count method. Phase 1 will be conducted to insure that HemoScreen is safely used for capillary self-testing by patient before initiating phase 2, where the HemoScreen is being sent home with the patients for self-measure at home.

Phase 1: Feasibility and usability of HemoScreen hematology analyzer for self-testing by cancer patients receiving chemo The aim of the study

* Comparison of capillary blood counts in patients, measured using the HemoScreen CBC analyzer versus laboratory measurements of venous blood counts, to indicate the reliability of results obtained from capillary self-testing by patients.
* To test the usability of HemoScreen by patients
* To evaluate the usability of HemoScreen by healthcare professionals
* Evaluate on training, before the initiation of phase 2
* To insure HemoScreen is safely used for capillary self-testing by patient before initiating phase 2

Study participants and study design This study aims to investigate the usability when performing blood testing during chemotherapy with HemoScreen CBC analyzer equipment, firstly for healthcare professionals and hereafter patients. Both patients and healthcare personnel will be instructed in using the equipment and will perform a self-test. The number of patients to be included is estimated to 10 and health professionals is 4-10. The duration of phase 1 will be approximately one month (September 2020).

Participants will be patients receiving chemo treatment for Breast Cancer at the Department of Clinical Oncology in Naestved, in the outpatient clinic and healthcare personnel at the Department of Clinical Oncology. The day before treatment, when the patients visit the hospital to have a standard venous blood test, patients will turn to the Department of Clinical Oncology to attend the study. The patients will receive introduction and intensive training regarding test procedure and operation of the device by a trained project nurse, and the nurse will draw a capillary blood test on the patient as part of the training. Hereafter, the patient will perform a self-test with HemoScreen. The nurse will furthermore instruct the patient how to upload the results to MY-SP.

The healthcare professionals who will test the usability of HemoScreen will also be instructed and trained the same way as the patients, and then perform a self-test with the HemoScreen CBC analyzer.

All participants, patients as well as healthcare personal will have a simple stepwise illustrative guide available when performing the self-test.

The study include a quantitative and a qualitative part. A quantitative comparison of capillary blood counts in patients, measured using the HemoScreen CBC analyzer versus laboratory measurements of venous blood counts, to indicate the reliability of results obtained from capillary self-testing by patients. Qualitative methods are used to explore the usability of HemoScreen for capillary blood counts when used by cancer patients and healthcare personal. Observations and semi-structured interviews will be conducted to identify eventually challenges and ensure that HemoScreen is suitable for self-testing by cancer patients. All participants enrolled in phase 1 of the study, will attend observation and interview. Observation and interview will be conducted at the hospital in connection to the training and self-test with HemoScreen.

Phase 2: Self-testing with HemoScreen in patients' home The aim of the study is to investigate

* How the patient experiences the use of HemoScreen for self-testing at home
* How the patients and relatives handle taking blood test in their own home in combination with a form (DBCG, Danish Brest Cancer Group, where the patients can register side effects)
* Explorative comparison of the result from capillary blood test with HemoScreen and laboratory results to see if HemoScreen results are reliable enough for clinical decisions

Study participants and study design This study aims to investigate the safety in letting patients perform blood tests at home during chemotherapy with HemoScreen equipment.

A trained nurse will identify patients at their first visit to the ward for outgoing patients. It will be patients receiving treatment for Breast Cancer at the Department of Clinical Oncology, Naestved. All participants enrolled in phase 2 of the study, will be trained and perform their first self-test with HemoScreen in the clinic, same procedure as phase 1. The subjective judgement of the patients' ability to conduct self-testing, will be used to secure its safe for the patient to be enrolled for self-testing at home. The patient is provided a simple stepwise illustrative guide on capillary blood test with HemoScreen, a guide the patient bring home together with the device. Patients can turn to a HOTline, answered by a trained project nurse, if the patient have doubts about the use of HemoScreen. Furthermore, the investigator will visit patients at home to observe proper use of the HemoScreen equipment.

The investigators define a success in the study if patients can use the HemoScreen equipment properly at home following the given instruction. Failure is defined as if patients have to call the HOTline, or are observed not to use the equipment properly at home.

The number of patients to be included will be 33, each patient will be included for approximately 16 weeks, as the patient receive chemotherapy. The duration of phase 2 will be approximately (September 2020- October 2022).

In phase 2, the patients will take blood test in a natural setting at home the day before the treatment. The patients will upload the data to MY-SP. The patient will be instructed how to do that as part of the training in using HemoScreen. The patients will also have blood samples taken at laboratorie as usual, and the result of the blood test from HemoScreen will not be used to prescribe the chemotherapy. All trial procedures are conducted in addition to standard care.

Furthermore, some of the patients recruited for home testing of HemoScreen, will participate an observational study as well as interview that aims to explore the experience of patients using HemoScreen at home. The observational study and interview will be conducted in the patient's home during the study period. It is necessary to conduct the studies at the patient's home to explore the use context. The estimated number of patients are 5-7, but inclusion will continue until data saturation is met.

Side effects and inconveniences There are no major side effects relate to using HemoScreen CBC analyzer. The finger prick test may cause transient soreness in the small area where the sample has been taken. There is also a risk of having to do more pricks to obtain enough blood to perform the test. However, the benefit to the patient by being able to perform blood counts in home exceeds by far the eventually disadvantage of a transient sore finger. The ability of cancer patients in chemotherapy to do blood counts at home would prevent wasted hospital journeys for the patient, and leave more time with relatives and family at home. When receiving chemo the patients have a reduced immune responds and are therefore at increased risk of getting an infection, therefore the less public transport and hospital visits the better. A further advantage is the ability to monitor the patient at home and reduce the risk of server side effects as neutropenia, anemia and thrombocytopenia complications. In addition, it would save hospital resources and least but not less involve the patient, and give them insight into own treatment.

The HemoScreen CBC analyzer is CE marked for point-of-care use. The device is not yet approved for use by patients.

Data The study (phase 1 and 2) collects all data according to the guidelines of Good Clinical Practice (GCP) for medical device studies. All data are pseudonymized, and all data are protected according to General Data Protection Regulation and Data protection Act.

The project has been reported to the Danish Data Protection Agency (Datatilsynet).

Economy Two HemoScreen devices used in phase 1 are bought and additional 8 devices will be leased. HemoScreen has no influence on the project and has no rights to data collected in the project.

Publications At least one scientific paper will be published upon completion of this study.

ELIGIBILITY:
Inclusion Criteria patients:

* Breast cancer patients receiving anti-cancer treatment at the Department of Oncology for outpatients
* 18 years old or more

Exclusion Criteria patients:

* Patients unable or unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and results
* Known bleeding disorders
* Bad circulation, if the patient cannot get enough blood drops to do the test
* Inability to give informed content due to mental capacity or language barrier

Inclusion Criteria Health-care professionals:

* Working at the Department of Oncology for outpatients
* 18 years old or more

Exclusion Criteria Health-care professionals:

* If unable or unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and result
* Known bleeding disorders
* Bad circulation, if the testperson cannot get enough blood drops to do the test
* Inability to give informed content

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The main study population will be patients diagnosed with breast cancer receiving anti-cancer treatment at the department of Oncology for outpatients. 10 patients in the first phase, testing the HemoScreen at the outpatient clinic only once, and 33 patients in the second phase testing in the outpatient clinic once as well as conducting self-testing at home during their anti-cancer treatment.
  A minor group of Health-care professionals from the Department of Oncology(between 5-10) will test the HemoScreen once in the ambulatory in the first phase.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The usability of PixCell HemoScreen for self-testing by cancer patients receiving chemo. | 16 weeks
  In phase 1 (ambulatory) and 2 (ambulatory and home): The patients will be observed when they perform self-testing in the ambulatory. The observer records in what order the different steps are conducted, and whether the different steps are performed correctly. The capability of each participant to perform self-testing will be evaluated. An overall capability score between 1-10 (1 low and 10 high performance) will be reported.
  The observation should identify the specific challenges in self-testing with HemoScreen and potential difficulties for the specific patient group. These observations will be reported.
  Furthermore, the patients will be interviewed about how they perceive their own performance at self-testing.
  In phase 2, a semistructured interview will be conducted in patients home to investigate how the patients experience self-testing with HemoScreen at home. Based on observations and qualitative date the usability of HemoScreen in home will be evaluated and reported.
Accuracy of capillary blood counts in self-testing with HemoScreen. Comparison of capillary self-test blood counts versus venous blood counts. | 16 weeks
  Comparison of capillary and venous blood counts will be performed to investigate the applicability of the capillary self-test performed by the patient. In phase 1 and 2 the patients will perform a capillary self-test with HemoScreen in ambulatory. Furthermore, a venous blood sample from the patient (drawn by nurse) will be analyzed at the Sysmex 9000 (standard procedure) and HemoScreen by nurse.
  In phase 2, further (approximately 5-6) capillary self-tests will be conducted by patients in patients own home. On the same day of capillary self-testing in home the patients will go to the hospital to have a venous blood sample drawn. The venous blood sample will be analyzed at Sysmex 9000 (standard procedure).
  Hematological components specified as measure 3, 4, 5 and 6 will be statistically compared with two sampled paired t-test, Deming regression and Pearson's correlation coefficient.
WBC (White blood cell) count | 16 weeks
  The total count of the white blood cells as well as differentiated count of white blood cells will be measured on HemoScreen as well as Sysmex 9000. The differentiated counts includes:
  Neutrophilocytes (10^9/L ) Lymphocytes (10^9/L ) Monocytes (10^9/L ) Eosinophilocytes (10^9/L ) Basophilocytes (10^9/L ) Deming regression, CV%, STD will be calculated to ensure the reliability of the results. The results will be evaluated specific to the lower range.
RBC (Red blood cell) count | 16 weeks
  The count of the red blood cells will be measured on HemoScreen as well as Sysmex 9000. The red blood cells is measured in unit: 10^9/L Deming regression, CV%, STD will be calculated to ensure the reliability of the results. The results will be evaluated specific to the lower range.
HGB (Hemoglobin) | 16 weeks
  Hemoglobin will be measured on HemoScreen as well as Sysmex 9000. Hemoglobin is measured in unit: mmol/L Deming regression, CV%, STD will be calculated to ensure the reliability of the results. The results will be evaluated specific to the lower range.
PLT (Platelets) count | 16 weeks
  The count of platelets will be analyzed on HemoScreen and Sysmex 9000. Platelets is measured in unit: 10^9/L Deming regression, CV%, STD will be calculated to ensure the reliability of the results. The results will be evaluated specific to the lower range.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henrik Holländer, MD, Principal Investigator — Zealand University hospital, Næstved
Locations (1):
- Zealand University Hospital, Oncology, Næstved, Denmark